CLINICAL TRIAL: NCT05129722
Title: Polydiuretic Therapy for Heart Failure With Preserved Ejection Fraction: A Pilot Trial
Brief Title: Polydiuretic Therapy for HFpEF, a Randomised Controlled Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties in recruitment at both sites.
Sponsor: The George Institute (Other)
Collaborators: Victor Chang Cardiac Research Institute (Unknown); St Vincent's Centre for Applied Medical Research (Unknown); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/PID02198
Record Dates: First submitted 2021-11-07; First posted 2021-11-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure with Preserved Ejection Fraction; HFpEF; Clinical Trial; SGLT2i; Sodium glucose co-transporter 2 inhibitor
MeSH Terms: interventions — Eplerenone; Bumetanide; empagliflozin

STUDY DESIGN:
Intervention Model Description: This pilot research project will be a multi-centre, double-blinded randomised control trial (1:1) of the use of a low dose combination polypill (bumetanide 0.5mg + eplerenone 25mg + empagliflozin 10mg) versus empagliflozin 10mg alone on top of their background therapy. There will be 15 patients per arm (n=30 across two sites).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomisation allocation will be blinded to all participants, physicians, and study team members, except an unblinded study statistician and study drug manufacturer. All individual, standard, and regulatory approved medications will be over-encapsulated and concealed by identical packaging, labelling, and administration scheduling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving low dose combination polydiuretic therapy (Experimental): This patient group will receive a low dose combination polydiuretic therapy treatment consisting of: bumetanide 0.5 mg (loop diuretic), eplerenone 25 mg (mineralocorticoid receptor antagonist) and empagliflozin 10mg (sodium-glucose co-transporter 2 inhibitor) daily on top of their background therapy.
  Interventions: Drug: Low dose combination polydiuretic therapy
- Comparator group receiving monotherapy empagliflozin (Active Comparator): This comparator patient group will receive empagliflozin 10mg (sodium-glucose co-transporter 2 inhibitor) daily on top of their background therapy.
  Interventions: Drug: Comparator monotherapy empagliflozin

INTERVENTIONS:
Drug: Low dose combination polydiuretic therapy — Low dose combination polydiuretic therapy treatment consists of:
  Loop diuretic bumetanide 0.5 mg Mineralocorticoid receptor antagonist eplerenone 25 mg Sodium-glucose co-transporter 2 inhibitor (SGLT2i): empagliflozin 10mg
  Other Names: Eplerenone (inspra), Bumetanide (Burinex) and Empagliflozin (jardiance)
  Arms: Patients receiving low dose combination polydiuretic therapy
Drug: Comparator monotherapy empagliflozin — Sodium-glucose co-transporter 2 inhibitor (SGLT2i): empagliflozin 10mg
  Other Names: Empagliflozin, Jardiance
  Arms: Comparator group receiving monotherapy empagliflozin

SUMMARY:
Heart Failure (HF) in Australia affects 1-2% of the population. Heart failure with preserved ejection fraction (HFpEF) refers to a syndrome of clinical heart failure without impairment of systolic cardiac function. HFpEF has few therapeutic agents that are proven to improve outcomes and it was only recently, the published EMPEROR-Preserved trial demonstrated that empagliflozin, a sodium-glucose cotransporter 2 inhibitor (SGLT2i) reduced composite outcome of heart failure hospitalisation and cardiovascular death by 21% among patients with HFpEF.[1] HFpEF therapies have traditionally aimed at providing symptomatic relief and treating coexisting illnesses.

This multi-centre randomised clinical trial aims to establish the feasibility of a fixed low dose combination polypill consisting of bumetanide 0.5 mg, eplerenone 25 mg, and empagliflozin 10 mg in patients with HFpEF compared against empagliflozin 10 mg monotherapy in patients with HFpEF.

Fixed dose combination low dose diuretics of this nature have not been rigorously studied in patients with HFpEF, and this study aims to help improve the treatment paradigm for this patient population.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) refers to a complex syndrome of clinical heart failure without impairment of systolic cardiac function. HFpEF accounts for more than half of patients with heart failure, and this prevalence continues to increase in population studies. Unlike Heart failure with reduced ejection fraction (HFrEF), there are few therapeutic agents that are proven to improve outcomes such as heart failure hospitalisation in this group. The recently published EMPEROR Preserved trial demonstrated that empagliflozin, a sodium-glucose cotransporter 2 inhibitor (SGLT2i), reduced the composite outcome of heart failure hospitalisation and cardiovascular death by 21% (95% CI: 10% to 31%) among patients with HFpEF. This was the first study to meet this clinical endpoint in HFpEF patients. In addition to reducing hospitalisation and CV death, additional therapies in HFpEF are aimed at providing symptomatic relief, through intravascular volume management with diuretics, and treating coexisting illnesses. However, patients may experience diuretic resistance that leads to lower efficacy of diuresis despite increasing doses; this, in turn, can lead to progression of renal dysfunction and other side effects.

Researchers and clinicians must develop strategies to help improve efficacy of diuresis and avoid diuretic resistance, which may be possible through the use of multiple diuretics at lower doses and including newer agents such as sodium-glucose cotransporter 2 (SGLT2) inhibitors.

This multi-centre, double-blinded, randomised (1:1), proof-of-concept, pilot trial aims to establish the feasibility of a fixed low dose combination polypill consisting of bumetanide 0.5 mg, eplerenone 25 mg, and empagliflozin 10 mg in patients with HFpEF compared against empagliflozin 10 mg monotherapy in patients with HFpEF. There will be 15 patients per arm (n=30 across two sites). The study will recruit patients from the community including cardiology clinics, primary care providers and will be undertaken in the Royal Prince Alfred (RPA) Cardiology Clinic and St Vincent's Hospital, Sydney, Australia Cardiology Clinic.

The primary implementation hypothesis for this study is that it is feasible to recruit 30 participants to this trial over 6 months and to complete 4 weeks of follow up, with adherence to the protocol and study related procedures (screening, randomisation, study drug allocation, follow-up procedures, and retention) in >/=80% of participants.

There are several secondary hypotheses including that the proposed polydiuretic, as compared to SGLT2i, empagliflozin monotherapy on top of usual care will: increase medication compliance, improve rates of optimal medical therapy, reduce N-terminal pro hormone BNP, improve New York Heart Association (NYHA) Class, reduce fluid overload, improve blood pressure, and body weight at 4 weeks alongside exploratory outcomes of change in their KCCQ. Additionally, the safety hypotheses include that patients will have no increase in Adverse events, Serious Adverse Events, or Adverse events of special interest.

Fixed dose combination low dose diuretics of this nature have not been rigorously studied in patients with HFpEF, and this study aims to help improve the treatment paradigm for this patient population. This combination of agents draws upon the existing nature of evidence based therapies used in HFpEF that target the kidney.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Adults ≥ 18 years old
3. Established diagnosis of NYHA Class II - IV heart failure with preserved ejection fraction, which has been present for at least 2 months
4. Left ventricular ejection fraction ≥50% on echocardiography within the last 12 months prior to study enrolment, and no previous echocardiogram with EF < 40% NB: Patients in which additional pharmacological or device therapy is contemplated, or should be considered, must not be enrolled until therapy has been optimised and is stable for ≥ 1 month.
5. NT-proBNP >300 pg/ml (or if hospitalised for heart failure within the previous 12 months, NT-proBNP ≥400 pg/ml) at enrolment. If concomitant atrial fibrillation at Visit 1, NT-proBNP must be ≥900 pg/ml (irrespective of history of heart failure hospitalisation)

Exclusion Criteria:

1. Known contraindication to bumetanide, eplerenone, or empagliflozin.
2. Concurrently prescribed prohibited medications which are mineralocorticoid receptor antagonists (Spironolactone and Eplerenone) and SGLT2i agents.
3. Symptomatic hypotension or systolic BP <95 mmHg at 2 out of 3 measurements at Visit 0
4. Current acute decompensated HF or hospitalisation due to decompensated HF <4 weeks prior to enrolment.
5. Myocardial infarction, unstable angina, stroke, or transient ischaemic attack (TIA) within 12 weeks prior to enrolment.
6. HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease or reduced EF < 50%
7. Symptomatic bradycardia or second or third-degree heart block without a pacemaker.
8. Evidence of secondary cause of hypertension e.g., renal artery stenosis; significant renal impairment (eGFR <50 ml/min/1.73 m2), raised serum potassium (above lab normal limit of 5.0 mEq/L).
9. Previous history of ketoacidosis
10. Women who are pregnant, breast feeding or of childbearing potential and are not using and do not plan to continue using medically acceptable form of contraception throughout the study (pharmacological or barrier methods).
11. Concomitant illness, physical impairment or mental condition which in the opinion of the study team / primary care physician could interfere with the conduct of the study including outcome assessment.
12. Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Participants in observational, natural history or epidemiological studies not involving an intervention are eligible.
13. Participant's responsible primary care or other responsible physician believes it is not appropriate for participant to participate in the study.
14. Inability or unwillingness to provide written informed consent.
15. Involvement in the planning and/or conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and compliance with study protocol (30 participants and 80% participant completion of study protocol) | 6 months
  Recruitment of 30 participants, with completion of study related procedures (screening, randomisation, study drug allocation, follow-up procedures, and retention over 4 weeks) in ≥ 80% of participants.

SECONDARY OUTCOMES:
NT-proBNP | 4 weeks
  Change in NT-proBNP (ng/L) from baseline to 4 weeks
NYHA Class | 4 weeks
  Change in NYHA Class (I-IV) from baseline to 4 weeks
6-minute Walk Test (6MWT) distance | 4 weeks
  Change in 6MWT distance (metres) from baseline to 4 weeks
Systolic and Diastolic Blood Pressure | 4 weeks
  Change in systolic and diastolic blood pressure (mmHg) from baseline to 4 weeks
Body Weight | 4 weeks
  Change in body weight from baseline to 4 weeks (Kg)
Haemoglobin A1c | 4 weeks
  Change in haemoglobin A1c (mmol//mol and %) from baseline to 4 weeks
Haemoglobin and haematocrit | 4 weeks
  Change in haemoglobin (g/L) and haematocrit from baseline to 4 weeks
Renal Function | 4 weeks
  Change in renal function measured by creatinine(umol/L) and estimated glomerular filtration rate (ml/min/1.73m2) from baseline to 4 weeks
Potassium | 4 weeks
  Change in blood potassium concentration (mmol/L) from baseline to 4 weeks
Total Diuretic Dose | 4 weeks
  Change in total diuretic dose from baseline to 4 weeks
Pill Burden | 4 weeks
  Number of pills taken during 4-week trial period

OTHER OUTCOMES:
Exploratory Endpoint | 4 weeks
  Changes in health-related quality of life measured by the Kansas City Cardiomyopathy Questionnaire from baseline to 4 weeks (scaled results 0-100 and higher number is reflective of a better outcome)
Incidence of Serious adverse events and Adverse events of special interest (safety and tolerability) | 4 weeks
  Incidence of treatment-emergent serious and special interest adverse events (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Arnott, Principal Investigator — The George Institute
Locations (2):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- [Background] Sahle BW, Owen AJ, Mutowo MP, Krum H, Reid CM. Prevalence of heart failure in Australia: a systematic review. BMC Cardiovasc Disord. 2016 Feb 6;16:32. doi: 10.1186/s12872-016-0208-4. PMID 26852410
- [Background] Bozkurt B, Coats AJ, Tsutsui H, Abdelhamid M, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Felker GM, Filippatos G, Fonarow GC, Fiuzat M, Gomez-Mesa JE, Heidenreich P, Imamura T, Januzzi J, Jankowska EA, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, SeferoviC P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal Definition and Classification of Heart Failure: A Report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure. J Card Fail. 2021 Apr;27(4):387-413. doi: 10.1016/j.cardfail.2021.01.022. Epub 2021 Mar 1. PMID 33663906